CLINICAL TRIAL: NCT05339282
Title: Necessity and Effectiveness of Empirical Antibiotic Use in Mild to Moderate Acute Inflammatory Gallbladder Disease; a Multicenter, Double-blind, Randomized, Placebo-controlled Trial
Brief Title: Effectiveness of Empirical Antibiotic Use in Mild to Moderate Acute Inflammatory Gallbladder Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Taeho Hong, Professor, Seoul St. Mary's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Seoul_S10
Record Dates: First submitted 2022-04-14; First posted 2022-04-21 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Cholecystitis, Acute
Keywords: empirical antibiotics; postoperative complication
MeSH Terms: conditions — Cholecystitis, Acute; Postoperative Complications | interventions — Cholecystectomy, Laparoscopic; Hematologic Tests; Blood Chemical Analysis; Urination; Blood Coagulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental group in acute cholecystitis (Experimental): inclusion criteria
  1. among patients with mild acute cholecystitis (grade I by Tokyo guidelines) or moderate acute cholecystitis without evidence of gallbladder perforation(grade II)
  2. cholecystitis with a thickness of 4 mm or more on gallbladder in preoperative imaging
  3. Gallbladder with surrounding organs due to gallbladder inflammation
  4. Patients over 19 years of age
  normal saline (Isotonic Sodium Chloride Injection Daihan(50mL/bag)) was used before surgery.
  Interventions: Procedure: Laparoscopic cholecystectomy
- The controled group in acute cholecystitis (Experimental): 1. among patients with mild acute cholecystitis (grade I by Tokyo guidelines) or moderate acute cholecystitis without evidence of gallbladder perforation(grade II)
  2. cholecystitis with a thickness of 4 mm or more on gallbladder in preoperative imaging
  3. Gallbladder with surrounding organs due to gallbladder inflammation
  4. Patients over 19 years of age
  First-generation cephalosporin (Cefazolin inj., 1g, Cefazolin sodium, Chong-geun-dang pharm.co.) was used before surgery.
  Interventions: Procedure: Laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: Laparoscopic cholecystectomy — Method of operation
  1. Surgery was started under general anesthesia
  2. A trocar of 10 mm was placed on the navel, 5 mm under the blade, and a 5 mm trocar was placed on the right upper abdomen.
  3. Pneumoperitoneum was performed using CO2 gas in the abdominal cavity.
  4. Dissection started from Calot's triangle, and the operation was performed by retrograde cholecystectomy.
  5. The excised gallbladder was placed in a laparoscopic pocket and extracted through the umbilicus.
  6. The trocar was removed, and the skin was sutured
  On the 1st day after surgery, hematology, blood chemistry, urine, blood clotting, and chest x-rays were performed. (Inspection and treatment were performed according to the current clinical pathway of gallbladder surgery)
  Other Names: hematology, blood chemistry, urine, blood clotting, and chest x-rays were performed

SUMMARY:
This clinical trial is an exploratory clinical trial that evaluates the necessity and effectiveness of empirical antibiotic use in mild and moderate acute inflammatory gallbladder diseases that require surgery, and the incidence of postoperative infection-related complications is compared.

DETAILED DESCRIPTION:
Cholecystectomy is the standard treatment for acute cholecystitis, accompanied by pain and fever due to acute inflammation in cholelithiasis patients. Empirical antibiotics are generally used to treat inflammation and prevent exacerbation before and after surgery. According to a previous study that confirmed the use of empirical antibiotics (JAMA. 2014;312(2):145-154. doi:10.1001/jama.2014.7586), the incidence of infectious complications was 15% in the group that used empirical antibiotics, and 15% of those who did not use empirical antibiotics The incidence of infectious complications in the group was 17%, confirming that there was no significant difference between the two groups. Based on these results, it was confirmed that the use of antibiotics after surgery was not clinically effective in reducing postoperative complications of infection.

However, there is a lack of objective research and evidence on the efficacy of empirical antibiotic use, and the use of antibiotics that have not been proven in practice may lead to the extension of hospital stay, waste of medical resources, and an increase in medical expenses. In addition, it can cause the occurrence of multidrug-resistant bacteria, which has been revived due to many problems recently, so caution is required in its use.

If the same anti-inflammatory effect and postoperative results can be obtained only through surgical treatment in mild and moderate acute inflammatory gallbladder disease, it is expected that the indiscriminate use of antibiotics will be reduced, and side effects thereof will be prevented. Therefore, this study intends to determine the effective and rational use of antibiotics through randomized clinical trials according to empirical antibiotics in laparoscopic surgery for patients with acute cholecystitis without evidence of systemic infection. In addition, a multicenter, double-blind, prospective, randomized, placebo-controlled clinical trial according to the use of empirical antibiotics has not been conducted in Korea so far, and thus clinical usefulness is expected to be great.

study population

1. Inclusion criteria

   * 19 years old or older - less than 70 years old
   * Those with mild (grade I by Tokyo guidelines) and severe (Grade Ⅱ) acute cholecystitis among the acute cholecystitis patient group
   * Cholecystitis with adhesions with surrounding organs due to gallbladder wall thickness of 4 mm or more or gallbladder inflammation
   * Those who voluntarily sign the written consent form after hearing and understanding the explanation of this clinical trial
2. Exclusion criteria

   * Those who are scheduled for elective gallbladder surgery (chronic cholecystitis, etc.)
   * Gallbladder disease that is not an inflammatory disease (GB cancer, GB polyp)
   * Pregnant or lactating women
   * A person who performs surgery at the same time due to other organ diseases
   * Those with immune suppression and bleeding tendency
   * Those who underwent percutaneous biliary drainage (PTGBD) before surgery
   * Those who require drainage tube installation during surgery
   * Those who are hypersensitive to cephalosproline antibiotics
   * Those who participated in other clinical trials within 3 months before screening
   * Other investigators who are judged inappropriate to participate in this clinical trial
3. Target number of subjects and calculation basis Since this study was a comparison with a reference drug, the number of subjects was calculated using a non-inferiority test. To calculate the number of study subjects, in the existing literature, the incidence of surgical site infection was 15% in the group using antibiotics and 17% in the group not using antibiotics. The difference value of the ratio between the two groups was 2% larger in the test group than in the control group, and the study subjects were calculated assuming 11%, the upper limit of the confidence interval between the two groups, as the non-inferiority margin. As a result, 166 subjects in each group are required, 10%. If the dropout rate is calculated, 185 per group, a total of 370 subjects, is required.

Study design

1. Design of clinical trials This clinical trial is an exploratory clinical trial evaluating the safety and effectiveness of using empirical antibiotics in mild and moderate acute inflammatory gallbladder disease requiring surgery. After determining whether the selection/exclusion criteria are suitable on the day of surgery, only suitable subjects are randomly assigned to the test group and control group in a 1:1 ratio. For the control group, the clinical investigational drug (Cefazolin 1g) was administered through an intravenous injection within 1 hour before the surgical site incision so that the concentration of antibiotics could be sufficiently maintained at the time of incision at the surgical site and the test group was administered with physiological saline without antibiotics do. Empirical antibiotics and saline are administered repeatedly at 24-hour intervals from the first dose until the patient is discharged.

   On the day of operation (OP day) and discharge, adverse reaction investigations, laboratory tests, and physical examinations for safety and efficacy evaluation are performed to evaluate the postoperative pain level and hospitalization period. One week after discharge, an outpatient visit is performed to evaluate adverse reactions, laboratory tests, and physical examinations to evaluate postoperative pain, the occurrence of postoperative infection-related complications, complications other than infection, and the need for additional procedures. In addition, when visiting the emergency room due to infection-related complications within a month after discharge, evaluate and compare the degree of postoperative pain, readmission, complications other than infection, and the need for additional procedures.
2. Method of subject registration and randomization Subjects who have listened to the explanation of this clinical trial and agreed to voluntarily participate in the trial will be given a subject identification code in the order in which they signed the consent form at the screening visit. Randomization is performed to ensure the scientific validity of clinical trials by ensuring that the subjectivity of the investigator is not involved in the assignment.

Block randomization is performed to divide the patients into 2 groups and allocate them in a 1:1 ratio for patients who satisfy the selection/exclusion criteria and agree to participate in the clinical trial. For randomization, a statistician independent of this clinical trial generates a randomization number using SAS ver.9.4 for Microsoft Windows (SAS Institute Inc, NC, Cary, USA) or higher and assigns them sequentially.

Method of operation

1. Surgery was started under general anesthesia
2. A trocar of 10 mm was placed on the navel, 5 mm under the blade, and 5 mm trocar was placed on the right upper abdomen.
3. Pneumoperitoneum was performed using CO2 gas in the abdominal cavity.

   * Double pressure through CO2 gas was maintained at 12mmHg / and 2L / min.
4. Dissection started from Calot's triangle, and the operation was performed by retrograde cholecystectomy.

   * The cystic duct was ligated with a 10mm clip, and the cystic artery was also ligated with a 10mm clip.
   * If the cystic duct was unstably ligated, ligation was performed through an end loop.
   * After ligation, the gallbladder was dissected from the liver.
5. Washed the surgical site.
6. The excised gallbladder was placed in a laparoscopic pocket and extracted through the umbilicus.
7. The trocar was removed, the skin was sutured, and the operation was completed.

characteristics of observational and clinical test

* Hematology tests: Hematocrit, Hemoglobin, Platelet, WBC & Differential count
* Blood coagulation test: PT INR, aPTT, BT
* Blood chemistry test: SGOT (AST), SGPT (ALT), alkaline phosphatase, γ-GTP, bilirubin (total / direct), fasting plasma glucose, BUN, creatinine, sodium, potassium, chloride, total protein, albumin, uric acid, CPK, LDH, CRP
* Imaging medical examination
* Postoperative hospital stay
* Check for infection.
* Check for leakage of bile.
* Surgery time and bleeding amount were described.
* Postoperative complications

Statistical analysis In the case of categorical variables for the length of stay, surgical time, and complication data obtained as secondary endpoints, n (%) was presented, and the ratio difference between the two groups was tested using Chi-square or Fisher's exact test. In addition, for continuous variables, the mean, standard deviation, median, minimum, and maximum values were presented. The normality test was performed to test with Student's t-test for normal distribution and the non-normal distribution Wilcoxon rank-sum test. The difference between the two groups would be tested. All statistical analyses would use SPSS version 21.0, and it would be judged that it was statistically significant below the significance level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. among patients with mild acute cholecystitis (grade I by Tokyo guidelines) or moderate acute cholecystitis without evidence of gallbladder perforation(grade II)
2. cholecystitis with a thickness of 4 mm or more on gallbladder in preoperative imaging
3. Gallbladder with surrounding organs due to gallbladder inflammation
4. Patients over 19 years of age, under 70 years of age

Exclusion Criteria:

1. patients with elective gallbladder surgery (chronic cholecystitis)
2. gallbladder disease not inflammatory disease (GB cancer, GB polyp)
3. pregnant women, patients under 18 years of age, over 70 years of age
4. patients with simultaneous surgery due to other organ diseases
5. immunosuppressed patients; liver transplant patients, kidney transplant patients, acquired immunodeficiency syndrome patients
6. patients with hemorrhagic tendency, or with hematologic diseases
7. Patients who underwent percutaneous cholecystectomy (PTGBD)

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Infectious Postoperative Complications | 30 days
  Incidence of infectious postoperative complications in patients who underwent a laparoscopic cholecystectomy due to grade I Tokyo guidelines for acute cholecystitis or grade II Tokyo guidelines for acute cholecystitis except the evidence of gallbladder perforation, with the first-generation cephalosporin and normal saline.

SECONDARY OUTCOMES:
Duration of hospitalization | Participants will be followed for the duration of hospital stay, an expected average of 2 days
  The duration between the operation day and the day of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Sung eun Park, MD, Study Director — The Catholic University of Korea
Locations (1):
- Department of HBP Surgery, Seoul St. Mary's hospital, Seoul, Seocho-gu, Banopo-dong, South Korea

IPD SHARING:
Plan to Share IPD: No